CLINICAL TRIAL: NCT00940121
Title: A Phase 1, Open-Label, Randomized, Parallel Dose Group Study to Assess the Pharmacokinetics of Mirabegron OCAS Formulations With Different Release Rates Versus IV Infusion in Healthy Volunteers
Brief Title: Pharmacokinetics of Oral Mirabegron With Different Release Rates Versus Intravenous (IV) Mirabegron
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 178-CL-076
Record Dates: First submitted 2009-07-13; First posted 2009-07-15 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2018-10

CONDITIONS: Healthy; Pharmacokinetics of Mirabegron
Keywords: oral administration; YM178; IV infusion; pharmacokinetics; mirabegron; Healthy volunteer subjects
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. mirabegron, low dose (Experimental): Oral mirabegron 25 mg
  Interventions: Drug: mirabegron
- 2. mirabegron, middle dose (Experimental): Oral mirabegron 50 mg
  Interventions: Drug: mirabegron
- 3. mirabegron, higher dose (Experimental): Oral mirabegron 100 mg
  Interventions: Drug: mirabegron

INTERVENTIONS:
Drug: mirabegron — oral tablet
  Other Names: YM178
Drug: mirabegron — IV solution
  Other Names: YM178

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of three doses of oral mirabegron formulations with three different release rates versus three doses of mirabegron administered intravenously; to study safety and side effects of the oral and IV doses of mirabegron.

DETAILED DESCRIPTION:
Subjects will be randomly assigned to one of three oral mirabegron doses and then randomly assigned to one of three oral mirabegron doses and then randomly assigned to one of six treatment sequences.

For all subjects the first treatment will be a reference IV dose. Treatments 2, 3, and 4 will be a random order of slow, fast and target release oral doses of mirabegron. Treatment 5 will be a target release dose of mirabegron from a different batch.

There will be at least 10 day washout between dose administrations.

ELIGIBILITY:
Inclusion Criteria:

* The subject must weigh at least 45 kg and have a body mass index (BMI) between 20.0 and 32.0 kg/m2
* The subject must have a normal or clinically nonsignificant 12 lead ECG as well as normal or clinically non-significant laboratory test results
* Female subjects must be post-menopausal (defined as at least 2 years without menses) surgically sterile, or practicing effective contraception, and will continue to use effective contraception during the study period. All females must be non-lactating, and should have a negative pregnancy test result
* The subject must have negative test results for drugs of abuse and alcohol screens
* The subject must have a good venous access in both arms

Exclusion Criteria:

* The subject has evidence of QTc interval >430 msec for male, >450 msec for female
* The subject has liver function test values (ALT, AST, or bilirubin) above the upper limit of normal
* The subject has a history or presence of psychiatric illness, serious active or recurrent infection
* The subject has a previous history of cancer other than basal cell carcinoma or Stage 1 squamous cell carcinoma that has not been in remission for at least 5 years
* The subject has donated or lost ≥ 450 mL blood within 56 days prior to study drug administration or has donated plasma within 7 days prior to study drug administration
* The subject has received or is anticipated to receive a prescription drug within 14 days (within 30 days for any long acting treatments such as depot formulations). Subject has taken any over-the-counter (OTC) medications, including complementary and alternative medicines (except for oral contraceptives and occasional use of acetaminophen of up to 2000 mg/day but not more than 4 days per week) within 14 days
* The subject has consumed alcohol, xanthine derivative-containing beverages/food (tea/chocolate), grapefruit juice, grapefruit-containing products or Seville oranges (e.g., bitter marmalade) within 48 hours before admission into the unit
* The subject has used tobacco-containing products and nicotine-containing products within 6 months
* The subject consumes more than 5 units of alcoholic beverages (one unit is 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits) per week, or has a history of substance abuse, drug addiction, or alcoholism within past 2 years
* The subject is known to have hepatitis or HIV-1 and/or HIV-2, or is positive for hepatitis A antibody IgM, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2009-04-30 (Actual); Primary Completion 2009-07-13 (Actual); Study Completion 2009-07-13 (Actual)

PRIMARY OUTCOMES:
Characterize the pharmacokinetic profile of 3 doses of oral mirabegron formulations with three different release rates vs. three doses of mirabegron administered intravenously | 2 months

SECONDARY OUTCOMES:
Assess the safety and tolerability of three doses of orally administered mirabegron formulated with three different release rates | 2 months
Assess the safety and tolerability of intravenously administered mirabegron | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (1):
- Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Background] Eltink C, Lee J, Schaddelee M, Zhang W, Kerbusch V, Meijer J, van Marle S, Grunenberg N, Kowalski D, Drogendijk T, Moy S, Iitsuka H, van Gelderen M, Matsushima H, Sawamoto T. Single dose pharmacokinetics and absolute bioavailability of mirabegron, a beta(3)-adrenoceptor agonist for treatment of overactive bladder. Int J Clin Pharmacol Ther. 2012 Nov;50(11):838-50. doi: 10.5414/CP201782. PMID 22943933